CLINICAL TRIAL: NCT01192399
Title: Phase II Clinical Study of Eculizumab (h5G1.1-mAb) in Hemolytic Paroxysmal Nocturnal Hemoglobinuria (PNH) Patients
Brief Title: Safety and Efficacy Study of Eculizumab in Paroxysmal Nocturnal Hemoglobinuria Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C07-001
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: Hemolytic Paroxysmal Nocturnal Hemoglobinuria; Eculizumab; PNH; Japan
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Eculizumab (Experimental): Eculizumab intravenous infusions every week x 4 doses, then 900 mg 1 week later for 1 dose, then 900 mg every 2 weeks for 4 doses
  Interventions: Biological: Eculizumab

INTERVENTIONS:
Biological: Eculizumab
  Other Names: Soliris

SUMMARY:
A study to assess the safety and efficacy of eculizumab in Japanese patients with hemolytic PNH.

DETAILED DESCRIPTION:
The objective of this study was to assess the safety and efficacy of eculizumab in Japanese patients with hemolytic PNH. In addition, the pharmacokinetics (PK) and pharmacodynamics (PD) of eculizumab in Japanese patients were assessed and compared to that of non-Japanese patients who had participated earlier studies of eculizumab treatment in hemolytic PNH.

ELIGIBILITY:
Inclusion Criteria:

* Japanese individuals at least 12 years of age
* Diagnosis of PNH > 6 months
* At least one transfusion in the past 2 years for anemia or anemia-related symptoms
* LDH level ≥ 1.5 x upper limit of normal within 12 weeks
* Presence of a glycosylphosphatidylinositol (GPI)-deficient red blood cell (RBC) clone (type III cells) by flow cytometry of ≥10%
* Negative serum pregnancy test for women of child-bearing potential

Exclusion Criteria:

* Platelet count < 30,000/µL
* Absolute neutrophil count ≤ 500/µL
* Known or suspected hereditary complement deficiency
* History of hematopoietic stem cell transplant
* History of meningococcal disease

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Squinto, PhD, Study Director — Alexion Pharmaceuticals, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kanakura Y, Ohyashiki K, Shichishima T, Okamoto S, Ando K, Ninomiya H, Kawaguchi T, Nakao S, Nakakuma H, Nishimura J, Kinoshita T, Bedrosian CL, Valentine ME, Khursigara G, Ozawa K, Omine M. Safety and efficacy of the terminal complement inhibitor eculizumab in Japanese patients with paroxysmal nocturnal hemoglobinuria: the AEGIS clinical trial. Int J Hematol. 2011 Jan;93(1):36-46. doi: 10.1007/s12185-010-0748-9. Epub 2011 Jan 12. PMID 21222185

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eculizumab
Started | 29
Completed | 27
Not Completed | 2
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Eculizumab
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (12.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 29
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 29

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lactate Dehydrogenase
Time Frame: Baseline, Week 12
Measure: Mean (Standard Error); unit: Units/Liter
Arm/Group | Eculizumab
Number analyzed (Participants) | 29
Units/Liter
  Baseline | 1845.1 (115.34)
  Week 12 | 398.7 (99.15)
  Change from Baseline at Week 12 | -1446.4 (138.68)
Statistical Analysis 1: Comparison: Eculizumab; Test type: Other; p < 0.0001, Sign test

2. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale Total Score
Description: The FACIT-Fatigue scale, Version 4.0, is a collection of quality of life questionnaires pertaining to the management of fatigue symptoms due to a chronic illness. The FACIT-Fatigue is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function over the preceding 7 days. Patients score each item on a 5-point scale: 0 (Not at all) to 4 (Very much). Total scores range from 0 to 52, with higher score indicating better quality of life.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Eculizumab
Number analyzed (Participants) | 29
units on a scale
  Baseline | 38.5 (1.88)
  Change from Baseline at Week 12 | 4.1 (2.25)

3. Secondary Outcome: Change From Baseline in Paroxysmal Nocturnal Hemoglobinuria (PNH) Red Blood Cell (RBC) Count
Time Frame: Baseline, Week 12
Measure: Mean (Standard Error); unit: cells x 10^12/L
Arm/Group | Eculizumab
Number analyzed (Participants) | 29
cells x 10^12/L
  Baseline | 1.3 (0.14)
  Week 12 | 1.8 (0.19)
  Change from Baseline at Week 12 | 0.5 (0.10)

4. Secondary Outcome: Number of Units of Packed Red Blood Cells (pRBCs) Transfused
Description: Comparison of number of units of pRBCs transfused in the 12 weeks prior to the first dose of eculizumab, and between baseline and 12 weeks after the first dose of eculizumab
Time Frame: 12 weeks pre-treatment, baseline, 12 weeks post-treatment
Measure: Mean (Standard Error); unit: Units
Arm/Group | Eculizumab
Number analyzed (Participants) | 29
Units
  12 Weeks Pre-Dose | 5.2 (1.04)
  12 Weeks Post-Dose | 1.5 (0.67)
  Difference Post - Pre | -3.7 (1.12)

5. Secondary Outcome: Change From Baseline in Lactate Dehydrogenase (LDH) Area Under the Curve (AUC)
Time Frame: Baseline to Week 12
Measure: Mean (Standard Error); unit: U/L x Day
Arm/Group | Eculizumab
Number analyzed (Participants) | 29
U/L x Day | -113540.5 (10539.33)

6. Secondary Outcome: Change From Baseline in Plasma Free Hemoglobin
Time Frame: Baseline, Week 12
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Eculizumab
Number analyzed (Participants) | 29
mg/dL
  Baseline | 22.6 (2.61)
  Change from Baseline at Week 12 | -19.8 (2.71)

7. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 Score (Global Health Status)
Description: The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) incorporates 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea and vomiting), a global health status scale, and a number of single items assessing additional symptoms commonly reported by cancer patients (dyspnoea, loss of appetite, insomnia, constipation and diarrhea) and perceived financial impact of the disease. All of the scales and single-item measures range in score from 0 to 100. For global health status, a high score represents a high quality of life.
Time Frame: Baseline, Week 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Eculizumab
Number analyzed (Participants) | 28
units on a scale | 8.9 (6.39)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the full study period (12 weeks).
Groups:
- Eculizumab: 600 mg of eculizumab as intravenous (IV) infusion once a week for 4 doses, followed by 900 mg eculizumab IV infusion 1 week later for 1 dose, then 900 mg eculizumab IV infusion every 2 weeks for 4 doses.
Arm/Group | Eculizumab
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=29)
Pyrexia (General disorders) | 1
C-Reactive Protein Increased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=29)
Anaemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 2
Tinnitis (Ear and labyrinth disorders) | 2
Conjunctival haemorrhage (Eye disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Chest discomfort (General disorders) | 2
Fatigue (General disorders) | 2
Pyrexia (General disorders) | 2
Nasopharyngitis (Infections and infestations) | 12
Blood alkaline phosphatase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Headache (Nervous system disorders) | 15
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes